CLINICAL TRIAL: NCT02586571
Title: Growth and Body Composition in Breastfed Infants - Study on Age of Introduction of Complementary Foods in Iceland
Acronym: IceAge2
Status: Completed | Type: Observational
Sponsor: University of Iceland (Other)
Collaborators: Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); University College, London (Other)
Responsible Party: Principal Investigator, Geir Gunnlaugsson, Professor, University of Iceland
Other Study IDs: IS-UI-IceAge2
Record Dates: First submitted 2015-10-04; First posted 2015-10-26 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Adiposity; Body Composition, Beneficial; Growth Acceleration
Keywords: Body Composition; Breast Feeding; Growth; Infant; Milk, Human; Nutritional Sciences; Weaning
MeSH Terms: conditions — Obesity; Glucocorticoid Receptor Deficiency; Breast Feeding | interventions — Lactation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples will be obtained from all infants at 5.5 and 12 months of age. Breast milk samples will be obtained from all mothers when the child is 5.5 months of age.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Exclusive Breastfeeding A: Mother/infant pairs with exclusive breastfeeding up to 6 months of age. Secondary outcome measure 2 (Metabolisable energy content of breast milk) measured in this group only.
  Interventions: Behavioral: Breastfeeding
- Exclusive Breastfeeding B: Mother/infant pairs with exclusive breastfeeding up to 6 months of age.
  Interventions: Behavioral: Breastfeeding
- Partial Breastfeeding: Mother/infant pairs with partial breastfeeding along with complementary foods at 6 months of age.
  Interventions: Behavioral: Breastfeeding

INTERVENTIONS:
Behavioral: Breastfeeding — Breastfeeding at 5.5 months of age (exclusive or partial)

SUMMARY:
The purpose of this prospective cohort study is to investigate breast-milk and breastfeeding among infants who are exclusively and partially breastfed at 6 months of age in terms of characteristics that are hypothesised to contribute to growth and development of body composition in infancy.

The scientific originality lies in the simultaneous sampling of multiple factors that are believed to contribute to growth and development of body composition in infancy, i.e. energy content of breast-milk, metabolism-regulating hormones in breast-milk, infant temperament and appetite. The selection of two predefined study groups, i.e. infants exclusively breastfed until 6 months of age and infants given complementary foods in addition to breast-milk from 3-4 months of age, gives the opportunity to describe, and perhaps up to some point compare, what now is described by the World Health Organization and in official Icelandic infant recommendations as "optimal feeding" and what studies have suggested is "common feeding" in many countries. The methods are carefully chosen, i.e. appropriate and non-invasive isotopes and validated questionnaires are used. To our knowledge, no study has reported breast-milk composition in exclusively vs. partially breastfed infants.

DETAILED DESCRIPTION:
At approximately 5 months of age, all infants in Iceland are invited to receive routine care (health checkup, immunization etc.) at the well-baby clinics at the primary health care centers in their neighbourhood. Nurses at well-baby clinics in and around Reykjavik cooperating with the study investigators screen all infants for eligibility according the eligibility criteria. Mothers of eligible infants receive oral and written information about the study and if interested, a written consent is obtained and study investigators are informed about the potential participant.

When the infant is around 5.5 months of age, the mother is contacted and a home visit by study investigators scheduled. In the home visit, more detailed information about the study is given and equipment for predose urine samples are given. The date for the first part of the study (day 0) is scheduled.

Day -1 and/or day 0: Mothers sample predose urine sample(s): 2x4 ml for group "Exclusive Breastfeeding A" and 1x2 ml for groups "Exclusive Breastfeeding B" and "Partial Breastfeeding".

Day 0 (home visit by investigators): Infant weighed, drinks 2.5 g/kg body weight + 1 g doubly labeled water or 0.7 g deuterium.

Mothers sample postdose urine samples: 6x4 ml for group "Exclusive Breastfeeding A" (days 1, 2, 3, 5, 6, 7) and 2x2 ml for the other groups (days 0+5 hours and day 2).

Mothers of infants in groups "Exclusive Breastfeeding B" and "Partial Breastfeeding" keep a 3-day weighed food record assessing their infants' diet including breast milk (by test weighing).

Day 7 (home visit by investigators): 2x10 ml breast milk samples (fore and hind milk) are obtained, questionnaires answered by mothers: background questionnaire, food frequency questionnaire on mother's habitual diet, the Baby Eating Behaviour Questionnaire (BEBQ) and the Infant Behaviour Questionnaire-Revised (IBQ-R).

At 9 months of age mothers keep a 3-day weighed food record assessing the infants' diet including breast milk if the infant is still breastfed (by test weighing).

At 12 months of age the primary outcome measure is assessed. Day -1 or day 0: Mothers sample predose urine sample: 1x2 ml. Day 0 (home visit by investigators): Infant weighed, drinks 1.2 g deuterium. Mothers sample postdose urine samples: 2x2 ml (days 0+5 hours and day 2). Mothers keep a 3-day weighed food record assessing their infants' diet including breast milk if the infant is still breastfed (by test weighing).

Mothers answer the Child Eating Behaviour Questionnaire (CEBQ).

ELIGIBILITY:
Inclusion Criteria:

* Icelandic mother
* Singleton birth
* Gestational age 37-42 weeks
* Birth weight >2500 g
* Living in Iceland until 12 months of age
* Only groups "Exclusive Breastfeeding A" and "Exclusive Breastfeeding B": Exclusively breastfed at 5.5 months of age (≤5 formula feedings and ≤5 water feedings since birth allowed)
* Only group "Partial Breastfeeding": Receiving at least 100 g / 100 ml of complementary foods (formula or solids) at 5.5 months of age

Exclusion Criteria:

* Diseases or defects likely to affect growth or body composition
* Not breastfed at 5.5 months of age

Ages: 5 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants receiving routine care at well-baby clinics at primary health care centers in and around Reykjavik, Iceland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Total body water measured by deuterium oxide | 12 months of age of child
  Total body water measured by deuterium oxide and used to determine fat-free mass

SECONDARY OUTCOMES:
Metabolisable energy content of breast milk measured using doubly labelled water | 5.5 months of age of child
  Measured using doubly labelled water (this outcome only measured in group labeled 'Exclusive Breastfeeding A')
Weight measured by infant scales | 0-12 months of age of child
  Weight measured by infant scales
Length measured by calibrated lengthboards | 0-12 months of age of child
  Length measured by calibrated lengthboards

OTHER OUTCOMES:
Infant eating behavior assessed using Baby Eating Behaviour Questionnaire (BEBQ) | 5.5 months of age of child
  Assessed using Baby Eating Behaviour Questionnaire (BEBQ)
Infant temperament assessed using the Infant Behaviour Questionnaire-Revised (IBQ-R) | 5.5 months of age of child
  Assessed using the Infant Behaviour Questionnaire-Revised (IBQ-R)
Leptin in breast milk | 5.5 months of age of child
  The metabolism-regulating hormone leptin measured in fore and hind milk samples
Ghrelin in breast milk | 5.5 months of age of child
  The metabolism-regulating hormone ghrelin measured in fore and hind milk samples
Cortisol in breast milk | 5.5 months of age of child
  The metabolism-regulating hormone cortisol measured in fore and hind milk samples
Infant eating behavior assessed using Child Eating Behaviour Questionnaire (CEBQ) | 12 months of age of child
  Assessed using Child Eating Behaviour Questionnaire (CEBQ)

CONTACTS AND LOCATIONS:
Overall Officials: Geir Gunnlaugsson, PhD, Principal Investigator — School of Social Sciences, University of Iceland; Inga Thorsdottir, PhD, Study Chair — School of Health Sciences, University of Iceland

REFERENCES:
- [Derived] Thorisdottir B, Odinsdottir T, Gunnlaugsson G, Eaton S, Fewtrell MS, Vazquez-Vazquez A, Kleinman RE, Thorsdottir I, Wells JC. Metabolizable Energy Content of Breastmilk Supports Normal Growth in Exclusively Breastfed Icelandic Infants to Age 6 Months. Am J Clin Nutr. 2023 Aug;118(2):468-475. doi: 10.1016/j.ajcnut.2023.06.005. Epub 2023 Jun 13. PMID 37369354
- [Derived] Petersen E, Thorisdottir B, Thorsdottir I, Gunnlaugsson G, Arohonka P, Erlund I, Gunnarsdottir I. Iodine status of breastfed infants and their mothers' breast milk iodine concentration. Matern Child Nutr. 2020 Jul;16(3):e12993. doi: 10.1111/mcn.12993. Epub 2020 Mar 11. PMID 32162412